CLINICAL TRIAL: NCT06549738
Title: Effects of Intermittent Pneumatic Compression Therapy on Tissue Volume, Pain, and Quality of Life in Women Living With Lipedema
Brief Title: Effects of Intermittent Pneumatic Compression Therapy on Tissue Volume, Pain, and Quality of Life in Lipedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lympha Press (Other)
Collaborators: Carolina Vein Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMM0089
Record Dates: First submitted 2024-07-10; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Lipedema
Keywords: lipedema; lipoedema
MeSH Terms: conditions — Lipedema | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled study planned for 50 women with lipedema with half (25) women in the Treatment group and half (25) women in the Control group. Both legs of all enrolled women will be studied for a total of 100 legs evaluated. All participants in the Treatment group will be supplied the Lympha Press Optimal Plus IPCD and the Lympha Pants™ garment to treat the lower body including the abdomen, pelvis, and buttocks (trunk) and the lower extremities. All participants in the study (Treatment and Controls) will receive compression leggings, and will be instructed to wear them daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Lympha Press Treatment. While the first IPCD treatment takes place in Visit 2, subjects will be educated on the use of the IPCD and the protocol they will follow for the home treatment phase. During the hour-long treatment session in the clinic, the pressure will be gradually increased per subject tolerance starting at 20 mm Hg. Subjects will be instructed to use the IPCD at home for 1-2 hours a day, with pressure set to patient tolerance (recommended setting of 45 mmHg).
  In addition to IPCD treatment, subjects will be provided compression leggings at Visit 1 and instructed to wear them daily during all waking hours until Visit 3.
  Interventions: Device: Intermittent pneumatic compression therapy
- Control (No Intervention): Subjects will be provided compression leggings at Visit 1 and instructed to wear them daily during all waking hours until Visit 3.

INTERVENTIONS:
Device: Intermittent pneumatic compression therapy — Lympha Press Optimal Plus is an advanced intermittent pneumatic compression therapy device. It is FDA cleared (K170658) for the indication of lipedema as well as for other indications for use.
  Other Names: Lympha Press; Lympha Press Optimal Plus; HCPCS code E0652; pneumatic compression; lymphedema pump
  Arms: Treatment

SUMMARY:
Lipedema is an inflammatory and painful disease of subcutaneous adipose tissue (SAT) in women that is associated with vein disease and lymphedema. There is controversy on whether there is edema in lipedema. This study seeks to determine: 1. Is there is edema in lipedema? 2. Can edema, lipedema subcutaneous adipose tissue (SAT), symptoms, and quality of life be improved by an advanced intermittent pneumatic compression device (IPCD)?

During the course of the study subjects will be seen three times in the clinic for assessment and measurements. All subjects will be provided a compression legging at the first clinic visit. Half of the subjects (the treatment group) will be provided and use an advanced intermittent pneumatic compression device with pants-type appliance that applies dynamic compression therapy to the abdomen, hips, buttocks, legs and feet, starting at the second visit, for 30 days at home, along with daytime use of the compression legging. The other half (the control group) will use the compression leggings only. At the third visit, final measurements will be obtained. The measurements in the study include volume measurements using tape measure and a scanner; body composition measurements (bioimpedance); ultrasound and biopsy of the skin; timed walking and gait measurements; and questionnaires about pain and quality of life. Deidentified (without names) patient medical records will be examined for information on vein disease, body mass index, weight, age, and stage of lipedema (any stage or type). After the third visit, results will be analyzed.

DETAILED DESCRIPTION:
Introduction Lipedema is a disease of loose connective (adipose) tissue that has no known cause or cure. One of the main features is an increased amount of abnormal fibrotic subcutaneous adipose tissue (SAT) deposited in the legs, pelvis, abdomen and/or arms of women.

Management options for lipedema focus on improving lymphatic flow, controlling edema (swelling), reducing pain or discomfort, and deep tissue therapy to try and reduce fibrosis. Intermittent pneumatic compression devices (IPCDs) are externally applied "pumps," that reduce leg swelling and improve pain and quality of life for patients with lipedema.

No study has demonstrated an improvement in fat volume (relative to total leg volume), fascia quality, and fibrosis of the leg after the use of IPCDs.

The goal of this study is to improve our understanding of lipedema tissue and how use of the IPCD, Lympha Press® Optimal Plus with Lympha Pants™ garments, may improve tissue volume, fluid, quality, quality of life, and pain levels in women with lipedema.

This is a randomized, controlled study of 50 women with lipedema with 25 women in the Treatment group and 25 women in the Control group. Women with lipedema will be recruited from women with lipedema who have had their vein disease treated. Women in this part of the study will therefore have only lipedema without active treatable vein disease. Both legs of all enrolled women will be studied for a total of 100 legs evaluated. All participants in the Treatment group will be supplied the Lympha Press Optimal Plus IPCD and the Lympha Pants™ garment to treat the lower body including the abdomen, pelvis, and buttocks (trunk) and the lower extremities. All participants in the study (Treatment and Controls) will receive compression leggings, and will be instructed to wear them daily.

Primary Aims

After use of Lympha Press® Lympha Pants™ for 30 days, changes will be assessed in:

1. Leg and abdominal tissue volume
2. Leg and abdominal fluid volume
3. Pain level
4. Quality of life

Secondary Aim 1

After use of the Lympha Press® Lympha Pants™ for 30 consecutive days, the following changes will be assessed:

1. Tissue microvasculature
2. Mobility

Secondary Aim 2

Assess the size and/or degree of insufficiency of the greater and lesser veins of the legs of women with lipedema.

Investigational Aims

After use of the Lympha Press® Lympha Pants™ for 30 consecutive days, the following changes will be assessed:

1. Hyaluronic acid and other GAG levels in the blood
2. GAG levels in adipose tissue
3. Percentage of leaky vessels in the skin
4. Tissue fascia quality
5. Tissue fibrosis

Hypotheses

Hypotheses for Primary Aims

Use of the Lympha Press® Optimal Plus with Lympha Pants™ for 30 consecutive days will:

1. Reduce size or volume of SAT measured by:

   1. Ultrasound assessment of adipose tissue depth
   2. Circumferential measurement every 10 cm from the ankle to the upper thigh using a measuring board. This will be done at the same time each day.
   3. Natural (smallest) waist with a vertical measurement to the umbilicus, and waist and hip circumferential measurements following WHO guidelines.
   4. Volumetric measurement (LymphaTech, Georgia) using a validated three-dimensional scanner handheld device.
   5. Caliper measurements under the umbilicus, on the anterior thigh and medial thigh as previously measured in women with lipedema.
2. Reduce trunk and leg fluid volume measured by bioimpedance analyses (BIA) (SoZo, Digital Health Platform, Impedimed Company, San Diego, California).
3. Reduce pain measured by a visual analogue scale.

3. Improve quality of life measured by the following two validated questionnaires:

1. RAND (Rand Healthcare, Rand.org) 36-Item Health Survey 1.0 (SF-36)
2. Lower extremity functional scale (LEFS)

Hypotheses for Secondary Aims Secondary Aim 1

Use of the Lympha Press® Lympha Pants™ for 30 consecutive days will:

Improve micro-vessel structure measured by:

1. Biopsy of the skin: Skin biopsies have previously shown that blood vessels in the dermis are oriented in a perpendicular manner to the plane of the skin suggestive of inflammation. These vessels may revert back to their normal orientation due to reduction of inflammation, fibrosis, and GAGs in the skin.
2. Thermography: We will assess changes in tissue microvasculature after use of the Lympha Press Optimal Plus with Lympha Pants by thermography photos (FLIR) of the legs and hypothesize a decrease in the overall number of visible vessels. The room temperature must be constant for repeat measurements. Non-thermogenic (regular) photos will also be taken in case body contours need to be assessed to determine locations of brighter spots in the photos representing dilated blood vessels.
3. Mobility: Women with lipedema very often have mobility limitations. We anticipate that women who initially have limited mobility will improve after using the Lympha Press Optimal Plus for 30 days at home. Mobility will be measured by:

   1. The "Timed up and Go (TUG)" test
   2. Quantitative assessment of their walk several times across a special walking mat (GAITRite) that records and analyzes the pattern of their footsteps.

Secondary Aim 2

Vein Disease - Chart Review Study: We hypothesize that there will be enlarged veins in women with lipedema with minimal venous insufficiency based on unpublished studies and previous anecdotal clinical assessments. In addition to data collected on veins in these women, we will collect body mass index, weight, age, and stage of lipedema (any stage or type). No protected health information will be collected.

Hypotheses for Investigational Aims

The use of Lympha Press Lympha Pants after 30 consecutive days will:

1. Improve tissue fascia quality: The integrity and quality of SAT superficial and deep fascia layers will be assessed by visual analogue scale analysis of ultrasound images by three independent reviewers. Images from a previous study will be used to create a 5-point scale of fascia quality which the reviewers will use to assess fascia quality from tissue ultrasounds obtained from our study subjects.
2. Decrease tissue fibrosis: SAT fibrosis will be measured by:

   1. Echogenicity of SAT and muscle.
   2. Tissue Rigidity Assessment

Subject Use of the Lympha Press Pump at Home The subjects will use the Lympha Press pump at home at least once a day for 30 days.

Day 30 Final Visit (+/- 2 days) After 30 consecutive days of daily home use of the Lympha Press Optimal Plus with Lympha Pants, legs will be assessed.

IPCD Treatment (one hour) Lympha Press Treatment. While IPCD treatment takes place, subjects will be educated on the use of the IPCD and the protocol they will follow for the home treatment phase. During the hour-long treatment session in the clinic, the pressure will be gradually increased per subject tolerance starting at 20 mm Hg.

Measures documented from the chart study including the venous duplex ultrasound exam

1. Age
2. Height
3. Weight
4. Surgical history
5. Medical history
6. Family history
7. Allergies
8. Vein reflux: sapheno-femoral junction, proximal GSV, GSV knee, GSV distal, sapheno-popliteal junction, superficial saphenous vein (SSV) proximal
9. Vein size: sapheno-femoral junction, proximal GSV, GSV knee, GSV distal, sapheno-popliteal junction, superficial saphenous vein (SSV) proximal
10. Treatment for the GSV or SSV
11. Clinical (C), Etiological (E), Anatomical (A), and Pathophysiological (P) classification of the veins

Expected outcomes of the study

Lipedema has no known cure and few treatment options are available. IPCDs have been used to manage this disease for years and have been shown to be a promising option for treatment. We anticipate the following outcomes:

1. Publication on venous disease in women with lipedema.
2. Publication on effects of the Lympha Press Optimal Plus Pump and Lympha Pants garments on:

   1. Tissue volume
   2. Pain
   3. Quality of life
   4. Mobility
3. Publication on the effect of the Lympha Press® Optimal Plus and Lympha Pants garments on fibrosis in lipedema adipose tissue.

Data management and statistical analysis Confidentiality of all subjects will be strictly protected. Each patient will have an assigned patient ID; no names or dates of birth will be included in the database. The information that makes the patient identifiable will only be available to the researchers handling the information and this information will be destroyed after 6 years.

Statistics Overarching Data Analyses Data will be collected on an excel spreadsheet and imported into GraphPad PRISM for statistical purposes and graphing. Data will only use subject numbers. Data from each visit such as volume, BIA, SAT thickness, VAS pain scores, caliper measurements, GAITrite and TUG data will be averaged for each data point and either described in the text of the publication or compared to other data points using paired t-tests or repeated measures ANOVA. Significance will be set at α<0.05.

RAND 36-Item Health Survey 1.0 Data from the RAND 36-Item Health Survey 1.0 will be input into an excel spreadsheet. The RAND 36-Item Health Survey 1.0 assesses eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

ELIGIBILITY:
Inclusion Criteria:

1. Females age 18 - 70 years.
2. Diagnosis of Stage 2-3 Type II-III lipedema
3. Patients with an IPCD must agree to wash off the pump over 30 days prior to the study starting.
4. Must have pain score with or without pressure in any lipedema area of 3 or more out of 11-point Likert visual analogue scale.
5. Able to maintain their current diet and exercise regimen for the 60-day study.
6. Must be ambulatory.
7. Must be willing to wear compression during the study. Compression is provided at no cost as part of the study.
8. Consistent eating plan with weight stability (within 10 lbs or usual weight fluctuation per the patient) over three months.
9. Must agree to not change their diet and exercise during the study.

Exclusion Criteria:

1. Inability to understand the purpose of the study and complete consent.
2. Bed bound, preventing assessment of activities of daily living like the rest of the population we are studying.
3. Contraindications to IPCD use:

   1. serious arterial insufficiency measured as a monophasic pulse wave by Doppler
   2. edema due to decompensated congestive heart failure by history - all patients with a diagnosis of CHF will be excluded for purpose of the study
   3. active phlebitis by physical exam
   4. active deep vein thrombosis by history
   5. localized wound infection by physical exam
   6. cellulitis by physical exam
4. Lymphedema with minimal to no lipedema.
5. Positive Stemmer sign on the feet.
6. Weight > 375 lbs. (170 kg) due to weight restriction on bioimpedance device.
7. Undergoing surgery during the time of the study.
8. Weight loss surgery within the past 18 months.
9. Use of diuretic medication.
10. Participation in another research study at the time of the study.
11. Use of immunosuppressant medications including Gleevec, diosmin, methotrexate, corticosteroids, Plaquenil or other. If they are on these medications, they must wean off for one month or not participate in this study.
12. Medical illness deemed significant by the PI.
13. Waist to hip ratio > 0.85.
14. Undergoing manual therapy of any kind including massage, physical therapy, occupational therapy, manual lymphatic drainage therapy, instrument assisted soft tissue therapy or other deep tissue therapy. Subjects must agree to stop all manual therapy for one month prior to participation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
ultrasound assessment of adipose tissue deposits | 30 days
  ultrasound of lower extremities and hips to assess fascia, echogenicity and depth. The integrity and quality of SAT superficial and deep fascia layers will be assessed by visual analogue scale analysis of ultrasound images by three independent reviewers. Images from a previous study will be used to create a 5-point scale of fascia quality(16, 23) which the reviewers will use to assess fascia quality from tissue ultrasounds obtained from our study subjects. SAT fibrosis will be measured by:
  1. Echogenicity of SAT and muscle.
  2. Tissue Rigidity Assessment
tissue volume assessed by tape measure | 30 days
  leg volume assessed by circumferential measurements every 10 cm to upper thigh using Jobst measuring board; waist measurements assessed with vertical measurement to the umbilicus and waist and hip circumferential measurements according to WHO guidelines
Volumetric measurement | 30 days
  Volumetric measurement of lower torso and legs using a validated handheld three dimensional scanning device (Lymphatech Company)
Volumetric measurements by caliper | 30 days
  caliper measurements under the umbilicus, on the anterior thigh and medial thighs previously measured in women with lipedema
Tissue/fluid assessment by bioimpedance analysis | 30 days
  Leg and trunk fluid volume measured by bioimpedance analyses
Pain measured using visual analog scale | 30 days
  Leg pain measured by Visual Analog Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Quality of life questionnaire | 30 days
  Quality of life measured by validated questionnaire RAND 36-item Health Survey 1.0 (SF-36)
Lower extremity functional scale (LEFS) | 30 days
  he Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The scale for each question is 0 - 4, with 0 = extreme difficulty and 4 = no difficulty. The lower the score the greater the disability.
  * The minimal detectable change is 9 scale points.
  * The minimal clinically important difference is 9 scale points.
  * % of maximal function = (LEFS score) / 80 * 10

SECONDARY OUTCOMES:
Skin biopsy- presence of perpendicularly oriented blood vessels | 30 days
  Assessment of improvement in microvascular structure by skin biopsy. : Skin biopsies have previously shown that blood vessels in the dermis of lipedema patients are oriented in a perpendicular manner indicative of inflammation. The percentage of perpendicularly oriented blood vessels in each biopsy sample will be counted.
Thermography | 30 days
  We will assess changes in tissue microvasculature after use of the Lympha Press Optimal Plus with Lympha Pants by thermography photos (FLIR) of the legs and hypothesize a decrease in the overall number of visible vessels. The room temperature must be constant for repeat measurements. Non-thermogenic (regular) photos will also be taken in case body contours need to be assessed to determine locations of brighter spots in the photos representing dilated blood vessels.
Improvement in mobility as measured by Timed Up and Go (TUG) test | 30 days
  Timed Up and Go test (TUG) measures the time in seconds it takes for the subject to rise from a sitting position, walk 10 feet at a normal pace, turn around, walk back to the chair and sit down. We anticipate that use of the Lympha Press Optimal Plus will reduce (in seconds) the time it takes each subject to perform this test.
Chart review - enlarged veins | 30 days
  We will review the patient's clinic medical records for presence or absence of enlarged veins. No protected health information will be retrieved.
Improvement in mobility as measured by the Gait-Rite device | 30 days
  The GAITRite® system automates measuring temporal (timing) and spatial (distance) gait parameters (temporal/spatial) and 8 levels of relative pressure. Measurements of each subject will be taken to determine if treatment with the Lympha Press Optimal Plus changes gait as measured in step length, stride length, step width and foot angle.
Chart review for vein disease | 30 days
  We will review the patients' clinic medical records for presence or absence of venous disease. No protected health information will be retrieved.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Herbst, MD, PhD, Study Chair — The Roxbury Institute; Lynda McHutchison, Principal Investigator — Carolina Vein Center
Locations (1):
- Carolina Vein Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herbst KL, Kahn LA, Iker E, Ehrlich C, Wright T, McHutchison L, Schwartz J, Sleigh M, Donahue PM, Lisson KH, Faris T, Miller J, Lontok E, Schwartz MS, Dean SM, Bartholomew JR, Armour P, Correa-Perez M, Pennings N, Wallace EL, Larson E. Standard of care for lipedema in the United States. Phlebology. 2021 Dec;36(10):779-796. doi: 10.1177/02683555211015887. Epub 2021 May 28. PMID 34049453
- [Background] Bast JH, Ahmed L, Engdahl R. Lipedema in patients after bariatric surgery. Surg Obes Relat Dis. 2016 Jun;12(5):1131-1132. doi: 10.1016/j.soard.2016.04.013. Epub 2016 Apr 14. No abstract available. PMID 27317598
- [Background] Pouwels S, Huisman S, Smelt HJM, Said M, Smulders JF. Lipoedema in patients after bariatric surgery: report of two cases and review of literature. Clin Obes. 2018 Apr;8(2):147-150. doi: 10.1111/cob.12239. Epub 2018 Jan 25. PMID 29372593
- [Background] Pouwels S, Smelt HJ, Said M, Smulders JF, Hoogbergen MM. Mobility Problems and Weight Regain by Misdiagnosed Lipoedema After Bariatric Surgery: Illustrating the Medical and Legal Aspects. Cureus. 2019 Aug 14;11(8):e5388. doi: 10.7759/cureus.5388. PMID 31620316
- [Background] Al-Ghadban S, Cromer W, Allen M, Ussery C, Badowski M, Harris D, Herbst KL. Dilated Blood and Lymphatic Microvessels, Angiogenesis, Increased Macrophages, and Adipocyte Hypertrophy in Lipedema Thigh Skin and Fat Tissue. J Obes. 2019 Mar 3;2019:8747461. doi: 10.1155/2019/8747461. eCollection 2019. PMID 30949365
- [Background] Pessentheiner AR, Ducasa GM, Gordts PLSM. Proteoglycans in Obesity-Associated Metabolic Dysfunction and Meta-Inflammation. Front Immunol. 2020 May 19;11:769. doi: 10.3389/fimmu.2020.00769. eCollection 2020. PMID 32508807
- [Background] Bates DO, Levick JR, Mortimer PS. Change in macromolecular composition of interstitial fluid from swollen arms after breast cancer treatment, and its implications. Clin Sci (Lond). 1993 Dec;85(6):737-46. doi: 10.1042/cs0850737. PMID 8287667
- [Background] Liu NF, Zhang LR. Changes of tissue fluid hyaluronan (hyaluronic acid) in peripheral lymphedema. Lymphology. 1998 Dec;31(4):173-9. PMID 9949388
- [Background] Szolnoky G, Borsos B, Barsony K, Balogh M, Kemeny L. Complete decongestive physiotherapy with and without pneumatic compression for treatment of lipedema: a pilot study. Lymphology. 2008 Mar;41(1):40-4. PMID 18581957
- [Background] Szolnoky G, Varga E, Varga M, Tuczai M, Dosa-Racz E, Kemeny L. Lymphedema treatment decreases pain intensity in lipedema. Lymphology. 2011 Dec;44(4):178-82. PMID 22458119
- [Background] Volkan-Yazici M, Yazici G, Esmer M. The Effects of Complex Decongestive Physiotherapy Applications on Lower Extremity Circumference and Volume in Patients with Lipedema. Lymphat Res Biol. 2021 Feb;19(1):111-114. doi: 10.1089/lrb.2020.0080. Epub 2020 Oct 30. PMID 33124947
- [Background] Volkan-Yazici M, Esmer M. Reducing Circumference and Volume in Upper Extremity Lipedema: The Role of Complex Decongestive Physiotherapy. Lymphat Res Biol. 2022 Feb;20(1):71-75. doi: 10.1089/lrb.2020.0128. Epub 2021 Apr 5. PMID 33798399
- [Background] Atan T, Bahar-Ozdemir Y. The Effects of Complete Decongestive Therapy or Intermittent Pneumatic Compression Therapy or Exercise Only in the Treatment of Severe Lipedema: A Randomized Controlled Trial. Lymphat Res Biol. 2021 Feb;19(1):86-95. doi: 10.1089/lrb.2020.0019. Epub 2020 Dec 9. PMID 33297826
- [Background] Lu IM, Weiler MJ, Frank ND, Jordi J, Dixon JB. Monitoring Leg Lymphedema Over the Course of Therapy Using an Infrared System. Lymphat Res Biol. 2020 Aug;18(4):333-339. doi: 10.1089/lrb.2019.0036. Epub 2019 Dec 3. PMID 31800362
- [Background] Ibarra M, Eekema A, Ussery C, Neuhardt D, Garby K, Herbst KL. Subcutaneous adipose tissue therapy reduces fat by dual X-ray absorptiometry scan and improves tissue structure by ultrasound in women with lipoedema and Dercum disease. Clin Obes. 2018 Dec;8(6):398-406. doi: 10.1111/cob.12281. Epub 2018 Sep 24. PMID 30248251
- [Background] Jenkinson C, Coulter A, Wright L. Short form 36 (SF36) health survey questionnaire: normative data for adults of working age. BMJ. 1993 May 29;306(6890):1437-40. doi: 10.1136/bmj.306.6890.1437. PMID 8518639
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Allen M, Schwartz M, Herbst KL. Interstitial Fluid in Lipedema and Control Skin. Womens Health Rep (New Rochelle). 2020 Oct 14;1(1):480-487. doi: 10.1089/whr.2020.0086. eCollection 2020. PMID 33786515
- [Background] Curri SB, Merlen JF. [Microvascular disorders of adipose tissue]. J Mal Vasc. 1986;11(3):303-9. French. PMID 3772261
- [Background] Forner-Cordero I, Perez-Pomares MV, Forner A, Ponce-Garrido AB, Munoz-Langa J. Prevalence of clinical manifestations and orthopedic alterations in patients with lipedema: A prospective cohort study. Lymphology. 2021;54(4):170-181. PMID 35073621
- [Background] Gold EW. The quantitative spectrophotometric estimation of total sulfated glycosaminoglycan levels. Formation of soluble alcian blue complexes. Biochim Biophys Acta. 1981 Apr 3;673(4):408-15. doi: 10.1016/0304-4165(81)90472-4. PMID 6784773
- [Background] Herbst KL, Ussery C, Eekema A. Pilot study: whole body manual subcutaneous adipose tissue (SAT) therapy improved pain and SAT structure in women with lipedema. Horm Mol Biol Clin Investig. 2017 Sep 20;33(2):/j/hmbci.2018.33.issue-2/hmbci-2017-0035/hmbci-2017-0035.xml. doi: 10.1515/hmbci-2017-0035. PMID 28930626
- [Background] Fiegler W. [Ultrasonic demonstration of lipomatous tissues and tumors (author's transl)]. Rofo. 1981 Feb;134(2):157-61. doi: 10.1055/s-2008-1056328. German. PMID 6452357
- [Background] Herbst KL, Coviello AD, Chang A, Boyle DL. Lipomatosis-associated inflammation and excess collagen may contribute to lower relative resting energy expenditure in women with adiposis dolorosa. Int J Obes (Lond). 2009 Sep;33(9):1031-8. doi: 10.1038/ijo.2009.119. Epub 2009 Jul 21. PMID 19621017
- [Background] Beltran K, Herbst KL. Differentiating lipedema and Dercum's disease. Int J Obes (Lond). 2017 Feb;41(2):240-245. doi: 10.1038/ijo.2016.205. Epub 2016 Nov 18. PMID 27857136
- [Background] Avraham T, Zampell JC, Yan A, Elhadad S, Weitman ES, Rockson SG, Bromberg J, Mehrara BJ. Th2 differentiation is necessary for soft tissue fibrosis and lymphatic dysfunction resulting from lymphedema. FASEB J. 2013 Mar;27(3):1114-26. doi: 10.1096/fj.12-222695. Epub 2012 Nov 27. PMID 23193171
- [Background] Reed RK, Townsley MI, Zhao Z, Ishibashi M, Laurent TC, Taylor AE. Lymphatic hyaluronan flux from skin increases during increased lymph flow induced by intravenous saline loading. Int J Microcirc Clin Exp. 1994 Jan-Apr;14(1-2):56-61. doi: 10.1159/000178207. PMID 7960445
- [Background] Reeves KD, Sit RW, Rabago DP. Dextrose Prolotherapy: A Narrative Review of Basic Science, Clinical Research, and Best Treatment Recommendations. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):783-823. doi: 10.1016/j.pmr.2016.06.001. PMID 27788902
- [Background] Crescenzi R, Marton A, Donahue PMC, Mahany HB, Lants SK, Wang P, Beckman JA, Donahue MJ, Titze J. Tissue Sodium Content is Elevated in the Skin and Subcutaneous Adipose Tissue in Women with Lipedema. Obesity (Silver Spring). 2018 Feb;26(2):310-317. doi: 10.1002/oby.22090. Epub 2017 Dec 27. PMID 29280322
- [Background] Tsai SW, Hsu YJ, Lee MC, Huang HE, Huang CC, Tung YT. Effects of dextrose prolotherapy on contusion-induced muscle injuries in mice. Int J Med Sci. 2018 Jul 30;15(11):1251-1259. doi: 10.7150/ijms.24170. eCollection 2018. PMID 30123064
- [Background] Herbst KL. Rare adipose disorders (RADs) masquerading as obesity. Acta Pharmacol Sin. 2012 Feb;33(2):155-72. doi: 10.1038/aps.2011.153. PMID 22301856
- [Background] Azma K, Mottaghi P, Hosseini A, Salek S, Bina R. Venous insufficiency after prolonged standing: Is joint hypermobility an important risk factor? Adv Biomed Res. 2015 May 11;4:98. doi: 10.4103/2277-9175.156666. eCollection 2015. PMID 26015924
- [Background] Child AH, Gordon KD, Sharpe P, Brice G, Ostergaard P, Jeffery S, Mortimer PS. Lipedema: an inherited condition. Am J Med Genet A. 2010 Apr;152A(4):970-6. doi: 10.1002/ajmg.a.33313. PMID 20358611
- [Background] Pascucci A, Lynch PJ. Lipedema with multiple lipomas. Dermatol Online J. 2010 Sep 15;16(9):4. PMID 20875325
- [Background] Michelini S, Chiurazzi P, Marino V, Dell'Orco D, Manara E, Baglivo M, Fiorentino A, Maltese PE, Pinelli M, Herbst KL, Dautaj A, Bertelli M. Aldo-Keto Reductase 1C1 (AKR1C1) as the First Mutated Gene in a Family with Nonsyndromic Primary Lipedema. Int J Mol Sci. 2020 Aug 29;21(17):6264. doi: 10.3390/ijms21176264. PMID 32872468
- [Background] Mendes AM, Madon RJ, Flint DJ. Effects of cortisol and progesterone on insulin binding and lipogenesis in adipocytes from normal and diabetic rats. J Endocrinol. 1985 Aug;106(2):225-31. doi: 10.1677/joe.0.1060225. PMID 3894560
- [Background] Paolacci S, Precone V, Acquaviva F, Chiurazzi P, Fulcheri E, Pinelli M, Buffelli F, Michelini S, Herbst KL, Unfer V, Bertelli M; GeneOb Project. Genetics of lipedema: new perspectives on genetic research and molecular diagnoses. Eur Rev Med Pharmacol Sci. 2019 Jul;23(13):5581-5594. doi: 10.26355/eurrev_201907_18292. PMID 31298310
- [Background] Fukaya E, Flores AM, Lindholm D, Gustafsson S, Zanetti D, Ingelsson E, Leeper NJ. Clinical and Genetic Determinants of Varicose Veins. Circulation. 2018 Dec 18;138(25):2869-2880. doi: 10.1161/CIRCULATIONAHA.118.035584. PMID 30566020
- [Background] Felmerer G, Stylianaki A, Hollmen M, Strobel P, Stepniewski A, Wang A, Frueh FS, Kim BS, Giovanoli P, Lindenblatt N, Gousopoulos E. Increased levels of VEGF-C and macrophage infiltration in lipedema patients without changes in lymphatic vascular morphology. Sci Rep. 2020 Jul 2;10(1):10947. doi: 10.1038/s41598-020-67987-3. PMID 32616854
- [Background] WOLD LE, HINES EA Jr, ALLEN EV. Lipedema of the legs; a syndrome characterized by fat legs and edema. Ann Intern Med. 1951 May;34(5):1243-50. doi: 10.7326/0003-4819-34-5-1243. No abstract available. PMID 14830102
- [Background] Dean SM, Valenti E, Hock K, Leffler J, Compston A, Abraham WT. The clinical characteristics of lower extremity lymphedema in 440 patients. J Vasc Surg Venous Lymphat Disord. 2020 Sep;8(5):851-859. doi: 10.1016/j.jvsv.2019.11.014. Epub 2020 Jan 25. PMID 31992537
- [Background] Forner-Cordero I, Olivan-Sasot P, Ruiz-Llorca C, Munoz-Langa J. Lymphoscintigraphic findings in patients with lipedema. Rev Esp Med Nucl Imagen Mol (Engl Ed). 2018 Nov-Dec;37(6):341-348. doi: 10.1016/j.remn.2018.06.008. Epub 2018 Aug 28. English, Spanish. PMID 30166264
- [Background] Felmerer G, Stylianaki A, Hagerling R, Wang A, Strobel P, Hollmen M, Lindenblatt N, Gousopoulos E. Adipose Tissue Hypertrophy, An Aberrant Biochemical Profile and Distinct Gene Expression in Lipedema. J Surg Res. 2020 Sep;253:294-303. doi: 10.1016/j.jss.2020.03.055. Epub 2020 May 11. PMID 32407981
- [Background] Bauer AT, von Lukowicz D, Lossagk K, Aitzetmueller M, Moog P, Cerny M, Erne H, Schmauss D, Duscher D, Machens HG. New Insights on Lipedema: The Enigmatic Disease of the Peripheral Fat. Plast Reconstr Surg. 2019 Dec;144(6):1475-1484. doi: 10.1097/PRS.0000000000006280. PMID 31764671
- [Background] Westergren-Thorsson G, Hedstrom U, Nybom A, Tykesson E, Ahrman E, Hornfelt M, Maccarana M, van Kuppevelt TH, Dellgren G, Wildt M, Zhou XH, Eriksson L, Bjermer L, Hallgren O. Increased deposition of glycosaminoglycans and altered structure of heparan sulfate in idiopathic pulmonary fibrosis. Int J Biochem Cell Biol. 2017 Feb;83:27-38. doi: 10.1016/j.biocel.2016.12.005. Epub 2016 Dec 11. PMID 27974233
- [Background] Ma W, Gil HJ, Escobedo N, Benito-Martin A, Ximenez-Embun P, Munoz J, Peinado H, Rockson SG, Oliver G. Platelet factor 4 is a biomarker for lymphatic-promoted disorders. JCI Insight. 2020 Jul 9;5(13):e135109. doi: 10.1172/jci.insight.135109. PMID 32525843
- [Background] Herbst KL, Hansen EA, Cobos Salinas LM, Wright TF, Larson EE, Schwartz JS. Survey Outcomes of Lipedema Reduction Surgery in the United States. Plast Reconstr Surg Glob Open. 2021 Apr 23;9(4):e3553. doi: 10.1097/GOX.0000000000003553. eCollection 2021 Apr. PMID 33912372
- [Background] Di Renzo L, Cinelli G, Romano L, Zomparelli S, Lou De Santis G, Nocerino P, Bigioni G, Arsini L, Cenname G, Pujia A, Chiricolo G, De Lorenzo A. Potential Effects of a Modified Mediterranean Diet on Body Composition in Lipoedema. Nutrients. 2021 Jan 25;13(2):358. doi: 10.3390/nu13020358. PMID 33504026
- [Background] Cannataro R, Michelini S, Ricolfi L, Caroleo MC, Gallelli L, De Sarro G, Onorato A, Cione E. Management of Lipedema with Ketogenic Diet: 22-Month Follow-Up. Life (Basel). 2021 Dec 15;11(12):1402. doi: 10.3390/life11121402. PMID 34947933
- [Background] Cornely ME, Hasenberg T, Cornely OA, Ure C, Hettenhausen C, Schmidt J. Persistent lipedema pain in patients after bariatric surgery: a case series of 13 patients. Surg Obes Relat Dis. 2022 May;18(5):628-633. doi: 10.1016/j.soard.2021.12.027. Epub 2022 Jan 7. PMID 35144895
- [Background] Muluk SC, Hirsch AT, Taffe EC. Pneumatic compression device treatment of lower extremity lymphedema elicits improved limb volume and patient-reported outcomes. Eur J Vasc Endovasc Surg. 2013 Oct;46(4):480-7. doi: 10.1016/j.ejvs.2013.07.012. Epub 2013 Aug 21. PMID 23973278
- [Background] Iverson RE, Pao VS. MOC-PS(SM) CME article: liposuction. Plast Reconstr Surg. 2008 Apr;121(4 Suppl):1-11. doi: 10.1097/01.prs.0000308480.33644.56. PMID 18379377
- [Background] Eliason AH, Seo YI, Murphy D, Beal C. Adiposis Dolorosa Pain Management. Fed Pract. 2019 Nov;36(11):529-533. PMID 31892777
- [Background] Sandhofer M, Hanke CW, Habbema L, Podda M, Rapprich S, Schmeller W, Herbst K, Anderhuber F, Pilsl U, Sattler G, Sandhofer M, Moosbauer W, Sattler S, Schauer P, Faulhaber J, Maier S, Barsch M, Mindt S, Halk AB. Prevention of Progression of Lipedema With Liposuction Using Tumescent Local Anesthesia: Results of an International Consensus Conference. Dermatol Surg. 2020 Feb;46(2):220-228. doi: 10.1097/DSS.0000000000002019. PMID 31356433
- [Background] Herbst KL. Subcutaneous Adipose Tissue Diseases: Dercum Disease, Lipedema, Familial Multiple Lipomatosis, and Madelung Disease. 2019 Dec 14. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK552156/ PMID 31895524
- [Background] Lurie F, Passman M, Meisner M, Dalsing M, Masuda E, Welch H, Bush RL, Blebea J, Carpentier PH, De Maeseneer M, Gasparis A, Labropoulos N, Marston WA, Rafetto J, Santiago F, Shortell C, Uhl JF, Urbanek T, van Rij A, Eklof B, Gloviczki P, Kistner R, Lawrence P, Moneta G, Padberg F, Perrin M, Wakefield T. The 2020 update of the CEAP classification system and reporting standards. J Vasc Surg Venous Lymphat Disord. 2020 May;8(3):342-352. doi: 10.1016/j.jvsv.2019.12.075. Epub 2020 Feb 27. PMID 32113854
- [Background] Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg. 2000 Jun;31(6):1307-12. doi: 10.1067/mva.2000.107094. PMID 10842165
- [Background] Vasquez MA, Rabe E, McLafferty RB, Shortell CK, Marston WA, Gillespie D, Meissner MH, Rutherford RB; American Venous Forum Ad Hoc Outcomes Working Group. Revision of the venous clinical severity score: venous outcomes consensus statement: special communication of the American Venous Forum Ad Hoc Outcomes Working Group. J Vasc Surg. 2010 Nov;52(5):1387-96. doi: 10.1016/j.jvs.2010.06.161. Epub 2010 Sep 27. PMID 20875713
- [Background] Launois R, Reboul-Marty J, Henry B. Construction and validation of a quality of life questionnaire in chronic lower limb venous insufficiency (CIVIQ). Qual Life Res. 1996 Dec;5(6):539-54. doi: 10.1007/BF00439228. PMID 8993100
- [Background] Bilney B, Morris M, Webster K. Concurrent related validity of the GAITRite walkway system for quantification of the spatial and temporal parameters of gait. Gait Posture. 2003 Feb;17(1):68-74. doi: 10.1016/s0966-6362(02)00053-x. PMID 12535728
- [Background] Leahy S, Toomey C, McCreesh K, O'Neill C, Jakeman P. Ultrasound measurement of subcutaneous adipose tissue thickness accurately predicts total and segmental body fat of young adults. Ultrasound Med Biol. 2012 Jan;38(1):28-34. doi: 10.1016/j.ultrasmedbio.2011.10.011. Epub 2011 Nov 21. PMID 22104525
- [Background] Maurins U, Hoffmann BH, Losch C, Jockel KH, Rabe E, Pannier F. Distribution and prevalence of reflux in the superficial and deep venous system in the general population--results from the Bonn Vein Study, Germany. J Vasc Surg. 2008 Sep;48(3):680-7. doi: 10.1016/j.jvs.2008.04.029. Epub 2008 Jun 30. PMID 18586443